CLINICAL TRIAL: NCT04002817
Title: Giant Cell Tumor of the Bone in Patients Under 15 Years Old: a Single Institution Case-series
Brief Title: Giant Cell Tumor of the Bone in Young Patients
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: Pediatric GCTB
Record Dates: First submitted 2019-06-25; First posted 2019-07-01 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2019-06

CONDITIONS: Giant Cell Tumor of Bone
MeSH Terms: conditions — Giant Cell Tumor of Bone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
single institution cases series review of histological and clinical data of young patient with Giant Cell Tumors

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients under 15 years old treated at Rizzoli Institute from 01 January 1982 to 31 December 2018.
2. Diagnosis of giant cell tumor of bone, aneurysmatic bone cysts with solid features and giant cell reparative granuloma.
3. Histological slides/formalin-fixed paraffin-embedded tissue tumor blocks from archive available to perform the histology analysis
4. Written informed consent prior to any study-specific analysis and/or data collection

Exclusion Criteria:

1. Patients with histological diagnosis different from diagnosis of giant cell tumor, aneurysmatic bone cysts with solid features, and giant cell reparative granuloma.
2. Patients with no available material for additional immunohistochemical and molecular analysis

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: young patients with giant cell tumor of bone
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
selection and review of 50 cases of young patients with Giant Cell Tumor of bone. | at baseline (Day0)
  Investigators will review all the medical records, radiological imaging, and histological slides of all cases in order to collect the largest pediatric series.

SECONDARY OUTCOMES:
analysis of H3F3A mutation expression on tissue tumor material | at baseline (Day0)
  In all cases with enough available material, immunohistochemistry will be performed on tumor tissue material. Histone 3.3 (H3.3) genes, and H3F3A mutation will be analyzed with immunohistochemistry and/or by allele specific-PCR analysis in order to confirm that the lesions are a giant cell tumors of bone occurring in a non-canonic age group (skeletally immature patients).

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

REFERENCES:
- [Result] Campanacci M, Baldini N, Boriani S, Sudanese A. Giant-cell tumor of bone. J Bone Joint Surg Am. 1987 Jan;69(1):106-14. PMID 3805057
- [Result] Al-Ibraheemi A, Inwards CY, Zreik RT, Wenger DE, Jenkins SM, Carter JM, Boland JM, Rose PS, Jin L, Oliveira AM, Fritchie KJ. Histologic Spectrum of Giant Cell Tumor (GCT) of Bone in Patients 18 Years of Age and Below: A Study of 63 Patients. Am J Surg Pathol. 2016 Dec;40(12):1702-1712. doi: 10.1097/PAS.0000000000000715. PMID 27526293
- [Result] Dahlin DC, Cupps RE, Johnson EW Jr. Giant-cell tumor: a study of 195 cases. Cancer. 1970 May;25(5):1061-70. doi: 10.1002/1097-0142(197005)25:53.0.co;2-e. No abstract available. PMID 4910256

DOCUMENTS (1):
  • Study Protocol (2019-04-03): https://cdn.clinicaltrials.gov/large-docs/17/NCT04002817/Prot_000.pdf